CLINICAL TRIAL: NCT02382757
Title: Changing Diabetes in Children (CDiC): Type 1 Diabetes in Economically Underprivileged Children in India
Brief Title: Changing Diabetes in Children
Acronym: CDiC
Status: Terminated | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3982; U1111-1149-2666 (Other: WHO)
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children
  Interventions: Drug: insulin human

INTERVENTIONS:
Drug: insulin human — Children will receive conventional treatment with human insulin according to standard medical practice.

SUMMARY:
This study is conducted in Asia. The primary objective of the CDiC programme is to improve access to comprehensive diabetes care among the children with diabetes from the economically underprivileged section of the population and to establish a registry for this group of children with type 1 diabetes in India.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with type 1 diabetes
* Parents/caretakers agree to participate in the study
* Child belongs to the below poverty line economic strata (Centre Director certifies economic status for inclusion in to the study)

Exclusion Criteria:

* Children with type 2 diabetes
* Children from higher economic status
* Those getting coverage under other government / private schemes

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with type 1 diabetes aged below 18 years will be included.
Sampling Method: Probability Sample
Enrollment: 3089 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Patient assessments: Number of days on insulin | After 40 months
Number of days with home blood glucose monitoring | After 40 months
HbA1c (glycosylated haemoglobin) | After 40 months
Number of episodes of ketoacidosis | After 40 months
Number of episodes of severe hypoglycaemia | After 40 months
Long-term complications | After 40 months

SECONDARY OUTCOMES:
Percentage of children with HbA1c equal to or below 8.0 | After 40 months
Percentage of children who died during the study | After 40 months
Percentage of children lost to follow-up | After 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Bangalore, India

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com